CLINICAL TRIAL: NCT04042220
Title: Effect of Glucocorticoids on the Outcome of Gamma Knife Radiosurgically Treated Patients With Brain Metastases During Immunotherapy - An Explorative Study
Brief Title: Glucocorticoids, Immunotherapy and Radiosurgery for Brain Metastases
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Josa M Frischer, MD, PhD, Principal Investigator, Medical University of Vienna
Other Study IDs: 1648/2019
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Glucocorticoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GK + IT: Gamma Knife and immunotherapy
- GK + IT + GC: Gamma Knife, immunotherapy and glucocorticoids
  Interventions: Drug: Glucocorticoids
- GK only: Gamma Knife without immunotherapy

INTERVENTIONS:
Drug: Glucocorticoids — Effect of glucocorticoids (which are often prescribed for cerebral edema) on clinical outcome
  Groups: GK + IT + GC

SUMMARY:
Background. Brain metastases are the most common intracranial tumor and occur in 20-40% of all oncological patients. The most common primary cancer in brain metastases is lung cancer, followed by melanoma, breast cancer, renal cancer and colorectal cancer. The incidence of brain metastases has been increasing but the occurrence of brain metastases is still associated with high morbidity and poor prognosis. The main treatment methods are stereotactic radiosurgery (SRS), microsurgical resection and whole brain irradiation (WBRT). The stereotactic Gamma Knife Radiosurgery (GKRS) is a non-invasive method, applying high dose radiation into an exact defined volume within the cranium, and thereby associated with significantly decreased neurotoxicity. It is the only treatment method for multiple disseminated and thereby non-resectable brain metastases. A novel treatment method of brain metastases is the combination of GKRS and systematic immunotherapy (IT), targeted therapy (TT) or chemotherapy, which showed significant improvements in survival. Furthermore, patients with brain metastases often develop cerebral edema, which is commonly treated with glucocorticoids to relieve the symptoms and decrease the fluid accumulation, but the long-term use was shown to be unfavorable due to various side effects. One of the potentially concerning side effect of glucocorticoids is the immunosuppressive properties. This raises the question of whether glucocorticoids might influence the effect of immunotherapy.

Aim. The aim of the study is to evaluate if the use of glucocorticoids before, during and after treatment with gamma knife radiosurgery and immunotherapy effect the overall survival in patients with brain metastases, in contrast to patients undergoing gamma knife radiosurgery and immunotherapy alone. In addition, the effect of glucocorticoids on progression-free survival and clinical outcome will be evaluated. For the evaluation of the modern oncological treatment, patients with gamma knife radiosurgery, receiving immunotherapy, will be compared to patients not receiving immunotherapy.

Patients and methods. The investigators plan to conduct a observational prospective preliminary study including about 200 radiosurgically treated patients with brain metastases. Patients will be included to our study, if they were diagnosed with one of two most common primary cancers (lung cancer or melanoma) and were treated with at least one Gamma Knife radiosurgical treatment for at least one brain metastasis. For the outcome evaluation of the different treatment options, a comprehensive database will be established. The study participations will not interfere with any clincally indicated therapeutic decisions and the study participants will not be exposed to any additional risks.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who were treated with Gamma Knife Radiosurgery for at least one or more brain metastases and diagnosed with one of two most common primary cancers (lung cancer or melanoma)
* Patients over 18 years and under 90 years
* Written, signed informed consent for study particaption after study explanation

Exclusion Criteria:

* Patients under 18 years
* Patients over 90 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included in our study, if they were diagnosed with one of two most common primary cancers (lung cancer or melanoma) and were treated with at least one Gamma Knife radiosurgical treatment for at least one brain metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | Through completion of the study, an average of 1 year
  Time from first Gamma Knife Radiosurgical Treatment

SECONDARY OUTCOMES:
New brain metastases | Through completion of the study, an average of half a year
  Time until new brain metastases
Clinical outcome according to Karnofsky Performance Status Scale (KPS) | Through completion of the study, an average of 1 year
  Clinical condition at last follow up according to KPS. The KPS uses steps of 10%. Patients with 100% are not affected by their disease in everday activities, whereas 0% equals death.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No